CLINICAL TRIAL: NCT00147693
Title: Systematic Care for Informal Caregivers of Dementia Patients: An Efficient Approach?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Prof.dr. M. Vernooij-Dassen, Scientific Institute for Quality of Healthcare (IQ Healthcare) and Alzheimer Centre Radboud University, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: SCAD; ZonMw grant no 945-04-152
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Dementia, Vascular; Dementia; Alzheimer Disease; Lewy Body Disease
Keywords: Dementia; Alzheimer Disease; Lewy-Body; Cost*; Community (dwelling); Caregiver(s); Institutionalization; Quality of life; Randomized Control Trail; Vascular dementia
MeSH Terms: conditions — Dementia, Vascular; Dementia; Alzheimer Disease; Lewy Body Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Diagnosis of caregivers' problems
Behavioral: Professional service: treatment of problems by counseling or practical support

SUMMARY:
The objective is to ascertain the potential efficiency of a systematic care programme for caregivers of dementia patients. The research questions are:

* What are the costs and benefits of the Systematic Care Programme - Dementia (SCP-Dementia), as compared with usual care?
* What are the effects on the quality of life of patients and informal caregivers (spouse, relative), as compared with usual care?

DETAILED DESCRIPTION:
A major challenge for future health care is the care for dementia patients and their informal caregivers. In usual care, the problems of caregivers often remain invisible until a crisis occurs. This inhibition is partly the result of informal caregivers paying scant attention to their own problems. Another reason is that professionals may not know how to support informal caregivers pro-actively (Van Hout et al., 2000). Therefore the family support programme (Bengtson, 1985: Vernooij et al., 2000) has been transformed into a Systematic Care Programme (SCP-Dementia). The reasons for choosing and studying the efficiency of this programme are the potential to diagnose and treat problems systematically, to cover a wide range of individual problems, its flexibility in connecting interventions to these problems, its suitability for pro-activity and the positive effects of the programme found in our previous study (Vernooij et al., 2000). To study its efficiency a cluster randomised controlled trial design will be used. Randomisation will take place in each of three participating regions. Professionals in the ambulatory mental health care services (psychologists and social psychiatric nurses) will be randomly assigned to either the intervention group or the control group before the recruitment of patients and informal caregivers. The study population consists of pairs of patients and their informal caregivers visiting the ambulatory mental health care service for the first time. The intervention is the training in SCP-Dementia and its subsequent use. SCP-Dementia consists of an assessment of the caregiver's sense of competence and suggestions on how to deal with deficiencies in competence. The follow-up period is one year. The primary outcome is patients´ admissions to nursing homes or residential homes. The secondary outcome is quality of life. Caregivers´ quality of life is assessed by sense of competence (SCQ), depression (CES-D) and physical quality of life (EuroQol). Patients´ quality of life by behavioral problems is assessed by the NPI-Q and the QOL-AD-Scale. The difference in proposed effect was based on previous research in which 14% of the patients in the intervention group and 28% in the control group were institutionalized (Vernooij-Dassen, 1993;1995). To detect a 50% reduction in institutionalization rates with 80% power at the two sided significance level of 0.05, 132 patient-caregiver dyads would be needed for each of the intervention and control arm. We inflated this sample size by a design effect of 1.15 to 152 dyads per trial arm to allow for correlation of dyads within the same cluster (i.e. professional), assuming an average cluster size of four and an intracluster correlation coefficient of 0.05. Assuming a 25% dropout rate of patient-caregiver dyads, the study needed an final enrolment of 190 dyads in each trial arm. The economic evaluation is a cost-effectiveness analysis regarding a societal perspective. In the economic evaluation both costs and effects will be monetarized and consequently will result in a net benefit.

ELIGIBILITY:
Inclusion Criteria:

* Pairs of patients and their informal caregivers visiting the ambulatory mental health care service for the first time and treated by the professionals participating in the study

Exclusion Criteria:

* Patients and caregivers not mastering the Dutch language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2005-06; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Patients admissions to nursing homes or residential homes. This outcome is the most important input for the estimation of cost differences between the intervention group and controls. | after one year follow-up period

SECONDARY OUTCOMES:
Secondary outcome for cost estimation is patient and caregiver related costs estimated by "Resource Utilisation in Dementia" (RUD), including time spent on caregiving, use of health care services by caregivers and patients and additional productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Myrra M Vernooij-Dassen, PhD, Principal Investigator — Coordinator Alzheimer Centre UMC Nijmegen
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Spijker A, Verhey F, Graff M, Grol R, Adang E, Wollersheim H, Vernooij-Dassen M. Systematic care for caregivers of people with dementia in the ambulatory mental health service: designing a multicentre, cluster, randomized, controlled trial. BMC Geriatr. 2009 Jun 7;9:21. doi: 10.1186/1471-2318-9-21. PMID 19500421